CLINICAL TRIAL: NCT00095173
Title: A Phase III, Multi-Center, Multi-National, Randomized Withdrawal Study to Evaluate the Safety and Efficacy of BMS-188667 in Children and Adolescents With Active Polyarticular Juvenile Rheumatoid Arthritis (JRA)
Brief Title: BMS-188667 in Children and Adolescents With Juvenile Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-033
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Abatacept (Active Comparator): Double Blind Period
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Double Blind Period
  Interventions: Drug: Placebo
- Abatacept - Open Label (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — IV infusions, IV, 10mg/kg body weight, every 4 weeks, 6 months (unless a disease flare discontinued the patient earlier).
  Other Names: Orencia
  Arms: Abatacept
Drug: Placebo — IV infusions, IV, N/A, every 4 weeks, 6 months.
  Arms: Placebo
Drug: Abatacept — Solution, intravenous, Approximately 10 mg/kg fixed dose, based on subject's body weight; 500 mg for subjects weighing < 60kg; 750 mg for subjects weighing 60 to 100 kg; and 1 gram for subjects weighing > 100 kg, monthly
  Other Names: Orencia
  Arms: Abatacept - Open Label

SUMMARY:
The primary purpose of the clinical research study is to assess the safety of treating children and juvenile subjects with BMS-188667 (Abatacept). In addition, the study will assess the effectiveness of BMS-188667 in reducing disease activity of Juvenile Rheumatoid Arthritis (JRA) or Juvenile Idiopathic Arthritis (JIA) as measured by the time to occurrence of disease flare.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Juvenile Rheumatoid Arthritis or Juvenile Idiopathic Arthritis;
* Current active arthritis;
* Failed treatment with at least one disease modifying anti-rheumatic drug (DMARD);
* Subjects must discontinue use of any DMARD other than methotrexate prior to the first dose of study medication

Exclusion Criteria:

* Presence of infection or history of frequent acute or chronic infections;
* Joint replacement surgery required during the study or history of surgery on more than 5 joints;
* Live vaccines within 3 months of the first dose of study medication;
* Unresolved serious bacterial infection or chronic bacterial infection;
* Subjects who currently have intermittent fever due to JRA/JIA, rheumatoid rash, hepato-splenomegaly, pleuritis, pericarditis, or macrophage activation syndrome.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2003-12; Primary Completion 2006-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (10):
  - Omaha, Nebraska
  - Livingston, New Jersey
  - New Hyde Park, New York
  - Valhalla, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Local Institution, Bregenz, Austria
- Brazil (3):
  - Local Institution, Botucatu
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- France (2):
  - Local Institution, Paris
  - Local Institution, Strasbourg
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Bremen
  - Local Institution, Halle
  - Local Institution, Hamburg
- Italy (6):
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Roma
  - Local Institution, Trieste
- Mexico (5):
  - Local Institution, Guadalajara
  - Local Institution, Mexico City
  - Local Institution, Monterrey
  - Local Institution, Puebla City
  - Local Institution, San Luis Potosí City
- Local Institution, Lima, Peru
- Local Institution, Lisbon, Portugal
- Spain (2):
  - Local Institution, A Coruña
  - Local Institution, Valencia
- Local Institution, Lausanne, Switzerland

REFERENCES:
- [Derived] Ruperto N, Lovell DJ, Berman A, Anton J, Viola DO, Lauwerys B, Rama ME, Bohnsack J, Breedt J, Fischbach M, Lutz T, Minden K, Ally M, Rubio-Perez N, Gervais E, Van Zyl R, Wong R, Askelson M, Martini A, Brunner HI; Pediatric Rheumatology Collaborative Study Group (PRCSG) and the Paediatric Rheumatology International Trials Organisation (PRINTO). Abatacept as Monotherapy and in Combination With Methotrexate in Patients With Juvenile Idiopathic Arthritis: Analysis of 2 Phase III Trials. J Rheumatol. 2023 Nov;50(11):1471-1480. doi: 10.3899/jrheum.2022-1320. Epub 2023 Jul 15. PMID 37453737
- [Derived] Brunner HI, Tzaribachev N, Louw I, Calvo Penades I, Avila-Zapata F, Horneff G, Foeldvari I, Kingsbury DJ, Paz Gastanaga ME, Wouters C, Breedt J, Wong R, Askelson M, Zhuo J, Martini A, Lovell DJ, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG) investigators. Long-Term Maintenance of Clinical Responses by Individual Patients With Polyarticular-Course Juvenile Idiopathic Arthritis Treated With Abatacept. Arthritis Care Res (Hoboken). 2023 Nov;75(11):2259-2266. doi: 10.1002/acr.25156. Epub 2023 Jun 22. PMID 37221146
- [Derived] Lim LSH, Lokku A, Pullenayegum E, Ringold S. Probability of Response in the First Sixteen Weeks After Starting Biologics: An Analysis of Juvenile Idiopathic Arthritis Biologics Trials. Arthritis Care Res (Hoboken). 2023 Jun;75(6):1238-1249. doi: 10.1002/acr.25003. Epub 2023 Jan 18. PMID 36651601
- [Derived] Ruperto N, Brunner HI, Tzaribachev N, Vega-Cornejo G, Louw I, Cimaz R, Dare J, Espada G, Faugier E, Ferrandiz M, Gerloni V, Quartier P, Silva CA, Wagner-Weiner L, Gandhi Y, Passarell J, Nys M, Wong R, Martini A, Lovell DJ; Pediatric Rheumatology Collaborative Study Group (PRCSG) and the Paediatric Rheumatology International Trials Organisation (PRINTO). Absence of Association Between Abatacept Exposure and Initial Infection in Patients With Juvenile Idiopathic Arthritis. J Rheumatol. 2021 Jul;48(7):1073-1081. doi: 10.3899/jrheum.200154. Epub 2021 Jan 15. PMID 33452173
- [Derived] Lovell DJ, Ruperto N, Mouy R, Paz E, Rubio-Perez N, Silva CA, Abud-Mendoza C, Burgos-Vargas R, Gerloni V, Melo-Gomes JA, Saad-Magalhaes C, Chavez-Corrales J, Huemer C, Kivitz A, Blanco FJ, Foeldvari I, Hofer M, Huppertz HI, Job Deslandre C, Minden K, Punaro M, Block AJ, Giannini EH, Martini A; Pediatric Rheumatology Collaborative Study Group and the Paediatric Rheumatology International Trials Organisation. Long-term safety, efficacy, and quality of life in patients with juvenile idiopathic arthritis treated with intravenous abatacept for up to seven years. Arthritis Rheumatol. 2015 Oct;67(10):2759-70. doi: 10.1002/art.39234. PMID 26097215
- [Derived] Ruperto N, Lovell DJ, Li T, Sztajnbok F, Goldenstein-Schainberg C, Scheinberg M, Penades IC, Fischbach M, Alcala JO, Hashkes PJ, Hom C, Jung L, Lepore L, Oliveira S, Wallace C, Alessio M, Quartier P, Cortis E, Eberhard A, Simonini G, Lemelle I, Chalom EC, Sigal LH, Block A, Covucci A, Nys M, Martini A, Giannini EH; Paediatric Rheumatology International Trials Organisation (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). Abatacept improves health-related quality of life, pain, sleep quality, and daily participation in subjects with juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1542-51. doi: 10.1002/acr.20283. Epub 2010 Jul 1. PMID 20597110
- [Derived] Ruperto N, Lovell DJ, Quartier P, Paz E, Rubio-Perez N, Silva CA, Abud-Mendoza C, Burgos-Vargas R, Gerloni V, Melo-Gomes JA, Saad-Magalhaes C, Chavez-Corrales J, Huemer C, Kivitz A, Blanco FJ, Foeldvari I, Hofer M, Horneff G, Huppertz HI, Job-Deslandre C, Loy A, Minden K, Punaro M, Nunez AF, Sigal LH, Block AJ, Nys M, Martini A, Giannini EH; Paediatric Rheumatology International Trials Organization and the Pediatric Rheumatology Collaborative Study Group. Long-term safety and efficacy of abatacept in children with juvenile idiopathic arthritis. Arthritis Rheum. 2010 Jun;62(6):1792-802. doi: 10.1002/art.27431. PMID 20191582
- [Derived] Ruperto N, Lovell DJ, Quartier P, Paz E, Rubio-Perez N, Silva CA, Abud-Mendoza C, Burgos-Vargas R, Gerloni V, Melo-Gomes JA, Saad-Magalhaes C, Sztajnbok F, Goldenstein-Schainberg C, Scheinberg M, Penades IC, Fischbach M, Orozco J, Hashkes PJ, Hom C, Jung L, Lepore L, Oliveira S, Wallace CA, Sigal LH, Block AJ, Covucci A, Martini A, Giannini EH; Paediatric Rheumatology INternational Trials Organization; Pediatric Rheumatology Collaborative Study Group. Abatacept in children with juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled withdrawal trial. Lancet. 2008 Aug 2;372(9636):383-91. doi: 10.1016/S0140-6736(08)60998-8. Epub 2008 Jul 14. PMID 18632147
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 214 enrolled; in Per A, 190 treated; 24 not treated due to screening failures.170 completed Per A, 123 responders qualified to enter Per B. One subject did not enter Per B; 122 responders were randomized, 60 abatacept and 62 placebo. 36 of 47 Per A non-responders re-entered at Per C. Protocol violation occurred; 5yr old participant.
Groups:
- Abatacept (All Participants in Period A): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every 2 weeks for 3 doses.
- Abatacept (Period B): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for 6 months or until they experienced a flare (Period B).
- Placebo (Period B): Placebo: Dextrose 5% in water (D5W) or normal saline (NS) IV infusion, once every 2 weeks for 3 doses, then monthly up to 6 months. Participants were seated or in supine position during infusion.
- Abatacept (Period A Non-Responders in Period C): Participants not eligible to continue into Period B but re-entered in Period C. Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every two weeks for three doses (Period A) or once a month for up to 5 years (Period C).
- Abatacept (Period C): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for up to 5 years.
- Placebo (Period B) to Abatacept (Period C): Participants from Period B Placebo group entering Period C. Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for up to 5 years.
Period: Open-Label Lead-In Phase (Period A)
Arm/Group | Abatacept (All Participants in Period A) | Abatacept (Period B) | Placebo (Period B) | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Started | 190 | 0 | 0 | 0 | 0 | 0
Completed | 170 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 17 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Phase (Period B)
Arm/Group | Abatacept (All Participants in Period A) | Abatacept (Period B) | Placebo (Period B) | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Started | 0 (All participants did not continue; responders entered Period B; non-responders re-entered Period C.) | 60 (123 responders from Period A qualified;122 entered and were randomized to abatacept and placebo.) | 62 (123 responders from Period A qualified;122 entered and were randomized to abatacept and placebo.) | 0 | 0 | 0
Completed | 0 | 49 | 31 | 0 | 0 | 0
Not Completed | 0 | 11 | 31 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 10 | 31 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Open-Label Extension Phase (Period C)
Arm/Group | Abatacept (All Participants in Period A) | Abatacept (Period B) | Placebo (Period B) | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Started | 0 | 0 | 0 | 36 (Participants were non-responders from Period A who re-entered in Period C.) | 58 (Includes 47 who completed Period B with no flare and 11 who discontinued Period B due to a flare) | 59 (Includes 33 who discontinued Period B due to a flare and 26 who completed Period B with no flare)
Completed | 0 | 0 | 0 | 13 | 29 | 27
Not Completed | 0 | 0 | 0 | 23 | 29 | 32
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 11 | 5 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 6 | 0
Not completed — No Longer Meets Study Criteria | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Poor/Non-Compliance | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 4 | 6 | 8

BASELINE CHARACTERISTICS:
Population: All treated participants in the Lead-In Phase (Period A)
Groups:
- Abatacept (All Participants in Period A): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes,once every 2 weeks for 3 doses, then monthly up to 6 months unless a disease flare discontinued the patient earlier.
Arm/Group | Abatacept (All Participants in Period A)
Number analyzed (Participants) | 190
Age, Continuous [Median (Full Range); unit: years] | 13.0 [5.0 to 17.0]
Gender [Count of Participants; unit: Participants]
  Female | 137
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Juvenile Rheumatoid Arthritis/Juvenile Idiopathic Arthritis (JRA/JIA) Disease Flare During Double-Blind Phase (Period B)
Description: Time to flare is defined as the elapsed number of days between the first dose date in Period B and the study day that disease flare is confirmed.
  All of the following criteria must be met to be defined as a flare:
  * > 30% worsening in at least 3 of the 6 JRA/JIA core response variables
  * > 30% improvement in not more than 1 of the 6 JRA/JIA core set variables
  * ≥ 2 cm of worsening must be present if the Physician or Parent Global Assessment is used to define flare
  * worsening in ≥ 2 joints must be present if the number of active joints or joints with limitation of motion is used to define flare based on changes in the surrogate marker, erythrocyte sedimentation rate (ESR)
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants
Measure: Median (Full Range); unit: months
Groups:
- Abatacept (Period B): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for 6 months or until they experienced a flare.
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
months | NA [NA to NA] — Fewer than 50% of the participants in the abatacept group experienced a flare, therefore the median time to flare is known to exceed 6 months, but cannot be estimated. | 6 [0.73 to 6.87]
Statistical Analysis 1: Comparison: Abatacept (Period B) vs Placebo (Period B); Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.16 to 0.59] — Abatacept over placebo

2. Secondary Outcome: Number of Participants With a Juvenile Rheumatoid Arthritis/Juvenile Idiopathic Arthritis (JRA/JIA) Disease With a Flare During Double-Blind Phase (Period B)
Description: All of the following criteria must be met to be defined as a flare:
  * > 30% worsening in at least 3 of the 6 JRA/JIA core response variables
  * > 30% improvement in not more than 1 of the 6 JRA/JIA core set variables
  * ≥ 2 cm of worsening must be present if the Physician or Parent Global Assessment is used to define flare
  * worsening in ≥ 2 joints must be present if the number of active joints or joints with limitation of motion is used to define flare based on changes in the surrogate marker, erythrocyte sedimentation rate (ESR)
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
participants | 12 | 33
Statistical Analysis 1: Comparison: Abatacept (Period B) vs Placebo (Period B); Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs During Open-Label Lead-In Phase (Period A)
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment.
  SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during the study and up to 28 days past study discontinuation. The select AEs were determined using the Medical Dictionary for Regulatory Activities (MedDRA, v14.1).
Time Frame: Period A (Day 1 to Day 113)
Population: All treated participants in Periods A
Measure: Number; unit: participants
Arm/Group | Abatacept (All Participants in Period A)
Number analyzed (Participants) | 190
participants
  SAE | 6
  Treatment-Related AE | 0
  All Deaths | 0
  Treatment-Related Deaths | 0
  Discontinuation of Study Drug due to AEs | 1

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs During Double-Blind Phase (Period B)
Description: as for outcome 3
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants in Periods B
Measure: Number; unit: participants
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
participants
  SAE | 0 | 2
  Treatment-Related AE | 0 | 0
  All Deaths | 0 | 0
  Treatment-Related Deaths | 0 | 0
  Discontinuation of Study Drug due to AEs | 0 | 0

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs During Open-Label Phase (Period C)
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during the study and up to 85 days past study discontinuation. The select AEs were determined using the Medical Dictionary for Regulatory Activities (MedDRA, v14.1).
Time Frame: Period C (Day 282 to end of study)
Population: All treated participants in Period C
Measure: Number; unit: participants
Groups:
- Abatacept (Period A Non-Responders in Period C): Participants not eligible to continue into Period B but re-entered in Period C. Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every two weeks for three doses (Period A) and once a month for up to 5 years (Period C).
Arm/Group | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Number analyzed (Participants) | 36 | 58 | 59
participants
  SAE | 9 | 9 | 12
  Treatment-Related AE | 2 | 4 | 3
  All Deaths | 0 | 0 | 1
  Treatment-Related Deaths | 0 | 0 | 0
  Discontinuation of Study Drug due to AEs | 1 | 2 | 3

6. Secondary Outcome: Median Percent Change From Baseline in JRA/JIA Core Set Variables During Double-Blind Phase (Period B)
Description: Percent change from baseline was calculated from the difference between post-baseline and baseline divided by baseline multiplied by 100 and reported as the range between 25th and 75th percentile, not full range; American College of Rheumatology (ACR) Pediatric 30 JRA/JIA core set variables include active joints, limited range of motion, physician global assessment of disease severity, parent global assessment of overall well-being, change in physical function as measured by the Childhood Health Assessment Questionnaire (CHAQ), erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP). Disease activity was assessed by the physician and parent on a 0-100 mm visual analog scale (VAS). Low values represent low severity of disease and good well-being whereas high values represent highly severe disease and very poor well-being.
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants in Period B
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
percentage change from baseline
  Active Joints | -20.9 [-92.0 to 17.86] | 50.00 [0.00 to 100.0]
  Joints with LOM | 0.00 [-45.5 to 0.00] | 50.00 [0.00 to 100.0]
  Physician Global Assessment | -29.8 [-86.3 to 22.48] | 55.95 [-31.3 to 250.0]
  Parent Global Assessment | -11.2 [-56.8 to 28.41] | 8.39 [-31.8 to 100.0]
  CHAQ Disability Index | 0.00 [-38.9 to 2.17] | 0.00 [-13.3 to 55.56]
  ESR | 0.00 [-20.7 to 50.00] | 20.50 [-14.3 to 92.00]
  CRP | 0.00 [-46.6 to 67.00] | 6.25 [-33.3 to 150.0]

7. Secondary Outcome: Median Percent Change From Baseline in JRA/JIA Core Set Variables During Open-Label Phase (Period C)
Description: Percent change from baseline was calculated from the difference between post-baseline and baseline divided by baseline multiplied by 100 and reported as the range between 25th and 75th percentile, not full range; American College of Rheumatology (ACR) Pediatric 30 JRA/JIA core set variables include active joints, limited range of motion, physician's global assessment of disease severity, parent global assessment of overall well-being, change in physical function as measured by the Childhood Health Assessment Questionnaire (CHAQ), erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP). Disease activity was assessed by the physician and parent on a 0-100 mm visual analog scale (VAS). Low values represent low severity of disease and good well-being whereas high values represent highly severe disease and very poor well-being.
Time Frame: Period C (Day 282 to end of study)
Population: All treated participants in Period C
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Number analyzed (Participants) | 36 | 58 | 59
percentage change from baseline
  Active Joints | -26.7 [-66.7 to 0.00] | -70.2 [-94.1 to -50.0] | -82.4 [-100 to -62.5]
  Joints with Limited Range of Motion | 0.00 [-33.3 to 36.67] | -50.0 [-75.0 to -27.3] | -71.4 [-86.2 to -23.1]
  Physician Global Assessment of Disease Severity | -31.9 [-50.0 to -9.33] | -75.0 [-91.3 to -52.3] | -81.8 [-91.4 to -64.3]
  Parent Global Assessment of Overall Well-Being | 1.96 [-19.6 to 26.67] | -62.7 [-93.8 to -27.5] | -63.9 [-84.2 to -38.8]
  CHAQ Disability Index | 14.14 [-16.7 to 100.0] | -56.7 [-81.8 to -18.2] | -45.5 [-75.0 to -12.5]
  ESR | 20.87 [-15.5 to 83.77] | -27.3 [-54.8 to 20.00] | -24.2 [-50.0 to 0.00]
  CRP | 0.00 [-31.6 to 43.68] | -33.8 [-84.4 to 54.84] | -27.8 [-75.0 to 11.11]

8. Secondary Outcome: Events of Special Interest During Open-Label Lead-In Phase (Period A), Including Infections, Peri-Infusional Adverse Events (AEs), Autoimmune Disorders and Malignancies
Description: The sponsor prospectively identified categories of AEs that may be associated with the use of immunomodulatory drugs including infections, peri-infusional AEs, autoimmune disorders, malignancies. Peri-infusional AEs are defined as those AEs of special interest occurring during the first 24 hours after the start of study drug infusion. Malignancies definitions were based on events in the MedDRA Maintenance and Support Services Organization (MSSO) malignancies Structured MedDRA Query (SMQ).Autoimmune disorders are in alignment with the pre-specified MedDRA codes of autoimmune disorders events of interest.
Time Frame: Period A (Day 1 to Day 113)
Population: All treated participants in Period A
Measure: Number; unit: participants
Arm/Group | Abatacept (All Participants in Period A)
Number analyzed (Participants) | 190
participants
  Infections and Infestations | 68
  Peri-Infusional AEs | 30
  Autoimmune Disorders | 2
  Malignancies | 0

9. Secondary Outcome: Events of Special Interest During Double-Blind Phase (Period B), Including Infections, Peri-Infusional Adverse Events (AEs), Autoimmune Disorders and Malignancies
Description: as for outcome 8
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants in Period B
Measure: Number; unit: participants
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
participants
  Infections and Infestations | 27 | 27
  Peri-Infusional AEs | 2 | 2
  Autoimmune Disorders | 0 | 0
  Malignancies | 0 | 0

10. Secondary Outcome: Events of Special Interest During Open-Label Phase (Period C), Including Infections, Peri-Infusional Adverse Events (AEs), Autoimmune Disorders and Malignancies
Description: as for outcome 8
Time Frame: Period C (Day 282 up to 56 days after the last dose of study medication)
Population: All treated participants in Period C
Measure: Number; unit: participants
Groups:
- Abatacept (All Participants in Period C): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for up to 5 years.
Arm/Group | Abatacept (All Participants in Period C)
Number analyzed (Participants) | 153
participants
  Infections and Infestations | 120
  Peri-Infusional AEs | 22
  Autoimmune Disorders | 7
  Malignancies | 1

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) Pediatric 30 (ACRP30), ACR Pediatric 50, ACR Pediatric 70, ACR Pediatric 90, and Inactive Disease Status Erythrocyte Sedimentation Rate (ESR) Response Rate
Description: The ACRP30 response criteria were defined as a ≥ 30% improvement over baseline in ESR. ACRP 50, 70, and 90 responses were defined similarly with 50%, 70%, and 90% improvements required, respectively.
Time Frame: Day 113, Day 282, and Day 2047
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Number analyzed (Participants) | 36 | 58 | 59
percentage of participants
  ACR Pediatric 30 (ESR) at Day 113 | 0 [NA to NA] — No participants with response | 100 [NA to NA] — Confidence interval not applicable if result is 100% | 100 [NA to NA] — Confidence interval not applicable if result is 100%
  ACR Pediatric 30 (ESR) at Day 282 | NA [NA to NA] — No participants in this group | 84.5 [75.2 to 93.8] | 67.8 [55.9 to 79.7]
  ACR Pediatric 30 (ESR) at Day 2047 | 69.2 [44.1 to 94.3] | 97.0 [91.1 to 100] | 86.7 [74.5 to 98.8]
  ACR Pediatric 50 (ESR) at Day 113 | 0 [NA to NA] — No participants with response | 65.5 [53.3 to 77.7] | 88.1 [79.9 to 96.4]
  ACR Pediatric 50 (ESR) at Day 282 | NA [NA to NA] — No participants in this group | 79.3 [68.9 to 89.7] | 52.5 [39.8 to 65.3]
  ACR Pediatric 50 (ESR) at Day 2047 | 69.2 [44.1 to 94.3] | 93.9 [85.8 to 100.0] | 80.0 [65.7 to 94.3]
  ACR Pediatric 70 (ESR) at Day 113 | 0 [NA to NA] — No participants with response | 37.9 [25.4 to 50.4] | 49.2 [36.4 to 61.9]
  ACR Pediatric 70 (ESR) at Day 282 | NA [NA to NA] — No participants in this group | 55.2 [42.4 to 68.0] | 30.5 [18.8 to 42.3]
  ACR Pediatric 70 (ESR) at Day 2047 | 53.8 [26.7 to 80.9] | 78.8 [64.8 to 92.7] | 63.3 [46.1 to 80.6]
  ACR Pediatric 90 (ESR) at Day 113 | 0 [NA to NA] — No participants with response | 17.2 [7.5 to 27.0] | 22.0 [11.5 to 32.6]
  ACR Pediatric 90 (ESR) at Day 282 | NA [NA to NA] — No participants in this group | 41.4 [28.7 to 54.1] | 15.3 [6.1 to 24.4]
  ACR Pediatric 90 (ESR) at Day 2047 | 38.5 [12.0 to 64.9] | 66.7 [50.6 to 82.8] | 40.0 [22.5 to 57.5]

12. Secondary Outcome: Number of Treated Participants With Marked Laboratory Abnormalities During Open-Label Lead-In Phase (Period A)
Description: Marked abnormalities were pre-defined as changes in lab tests that occurred after drug infusion and were reported relative to the normal range for each analyte. Hemoglobin, 11.6-14.8 grams per deciliter (g/dL);Hematocrit, 36.0-50.0 percent;Erythrocytes, 3.80-5.10x10*6 cells per microliter (c/uL);Platelets, 140-44 cells per liter (c/L);Leukocytes, 4.00-12.50 c/uL;Absolute Neutrophils + Bands, if <1.00x10^3 c/uL;Absolute Lymphocytes, if <0.72x10^3 or >7.50x10^3 c/uL;Absolute Eosinophils, if >0.750X10^3 c/uL;Alanine Aminotransferase, 0-40 units per liter (U/L);G-Glutamyl Transferase, 0-60 U/L;Bilirubin, 0.1-1.2 milligrams per deciliter (mg/dL);Blood Urea Nitrogen, 5.9-26.0 mg/dL;Creatinine, 0.50-1.50 mg/dL;Serum Potassium, 3.5-5.5 milliequivalents per liter (mEq/L);Serum Glucose, 65-99 mg/dL;Fasting Serum Glucose, 65-99 mg/dL;Total Protein, 6.0-8.5 g/dL;Albumin, 3.5-5.5 g/dL;Urine Protein, >=4;Urine Glucose, >=4;Urine Blood, >=4;Urine Red Blood Cells >=4;Urine White Blood Cells, >=4.
Time Frame: Period A (Day 1 to Day 113)
Population: All treated participants in Period C evaluated for a specific analyte.
Measure: Number; unit: participants
Groups:
- Abatacept (All Participants in Period A): Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every two weeks for three doses.
Arm/Group | Abatacept (All Participants in Period A)
Number analyzed (Participants) | 190
participants
  Hemoglobin (Low) n=189 | 2
  Hematocrit (Low) n=189 | 2
  Erythrocytes (Low) n=189 | 1
  Platelets (Low) n=189 | 1
  Platelet Count (High) n=189 | 2
  Leukocytes (Low) n=189 | 9
  Leukocytes (High) n=189 | 10
  Absolute Neutrophils + Bands (Low) n=189 | 5
  Absolute Lymphocytes (Low) n=189 | 9
  Absolute Eosinophils (High) n=189 | 16
  Alanine Aminotransferase (ALT, High) n=190 | 2
  G-Glutamyl Transferase (GGT, High) n=190 | 1
  Bilirubin (Total, High) n=190 | 1
  Blood Urea Nitrogen (High) n=190 | 6
  Creatinine (High) n=190 | 12
  Potassium (High) n=190 | 4
  Serum Glucose (Low) n=190 | 26
  Serum Glucose (High) n=190 | 2
  Fasting Serum Glucose (High) n=109 | 1
  Total Protein (High) n=190 | 2
  Albumin (Low) n=190 | 2
  Urine Protein (High) n=190 | 12
  Urine Glucose (High) n=190 | 1
  Urine Blood (High) n=190 | 23
  Urine White Blood Cells (High) n=75 | 9
  Urine Red Blood Cells (High) n=75 | 25

13. Secondary Outcome: Number of Treated Participants With Marked Laboratory Abnormalities During Double-Blind Phase (Period B)
Description: Marked abnormalities were pre-defined as changes in lab tests that occurred after drug infusion and were reported relative to the normal range for each analyte. Hemoglobin, 11.6-14.8 grams per deciliter (g/dL);Hematocrit, 36.0-50.0 percent;Erythrocytes, 3.80-5.10x10*6 cells per microliter (c/uL);Platelets, 140-44 cells per liter (c/L);Leukocytes, 4.00-12.50 c/uL;Absolute Neutrophils + Bands, if <1.00x10^3 c/uL;Absolute Lymphocytes, if <0.72x10^3 or >7.50x10^3 c/uL;Absolute Eosinophils, if >0.750X10^3 c/uL;Aspartate Aminotransferase, 0-40 units per liter (U/L); Alanine Aminotransferase, 0-40 U/L;Blood Urea Nitrogen, 5.9-26.0 mg/dL;Serum Sodium, 135-148 milliequivalents per liter (mEq/L);Serum Potassium, 3.5-5.5 mEq/L;Serum Glucose, 65-99 mg/dL;Fasting Serum Glucose, 65-99 mg/dL;Urine Protein, >=4;Urine Blood, >=4;Urine Red Blood Cells >=4;Urine White Blood Cells, >=4.
Time Frame: Period B (Day 113 to Day 282)
Population: All treated participants in Period B evaluated for a specific analyte.
Measure: Number; unit: participants
Arm/Group | Abatacept (Period B) | Placebo (Period B)
Number analyzed (Participants) | 60 | 62
participants
  Hemoglobin (Low) n=60, 61 | 1 | 1
  Hematocrit (Low) n=60, 61 | 1 | 1
  Erythrocytes (Low) n=60, 61 | 0 | 1
  Platelets (Low) n-60, 61 | 4 | 0
  Platelets (High) n=189 | 0 | 1
  Leukocytes (Low) n=60, 61 | 1 | 1
  Leukocytes (High) n=60, 61 | 1 | 2
  Absolute Neutrophils + Bands (Low) n=60, 62 | 0 | 1
  Absolute Lymphocytes (Low) n=60, 62 | 2 | 3
  Absolute Eosinophils (High) n=60, 62 | 6 | 4
  Aspartate Aminotransferase (AST, High) n=60, 62 | 1 | 0
  Alanine Aminotransferase (ALT, High) n=60, 62 | 1 | 0
  Blood Urea Nitrogen (High) n=60, 62 | 1 | 1
  Serum Sodium (Low) n=60, 62 | 0 | 1
  Serum Potassium (High) n=60, 62 | 2 | 0
  Serum Glucose (Low) n=60, 62 | 4 | 5
  Serum Glucose (High) n=60, 62 | 0 | 1
  Fasting Serum Glucose (High) n=60, 62 | 1 | 1
  Urine Protein (High) n=62 | 2 | 2
  Urine Blood (High) n=60, 62 | 12 | 6
  Urine White Blood Cells (High) n=24, 20 | 5 | 2
  Urine Red Blood Cells (High) n=24, 20 | 6 | 4

14. Secondary Outcome: Number of Treated Participants With Marked Laboratory Abnormalities During Open-Label Phase (Period C)
Description: Marked abnormalities were pre-defined as changes in lab tests after drug infusion and relative to normal range. Hemoglobin,11.6-14.8grams per deciliter(g/dL);Hematocrit,36.0-50.0 percent;Erythrocytes,3.80-5.10x10*6 cells per microliter(c/uL);Platelets,140-44 cells per liter(c/L);Leukocytes,4.00-12.50c/uL;Absolute(Abs)Neutrophils+Bands,<1.00x10^3 c/uL;Abs Lymphocytes,<0.72x10^3 or>7.50x10^3 c/uL;Abs Eosinophils,>0.750X10^3 c/uL;Alkaline Phosphatase,0-40 units per liter(U/L);Aspartate Aminotransferase,0-40 U/L;Alanine Aminotransferase,0-40U/L;G-Glutamyl Transferase,0-60 U/L;Bilirubin, 0.1-1.2 milligrams per deciliter(mg/dL);Blood Urea Nitrogen,5.9-26.0 mg/dL;Creatinine, 0.50-1.50mg/dL;Inorganic Phosphorus,2.8-6.2 U/L;Serum Potassium,3.5-5.5 milliequivalents per liter(mEq/L);Serum Glucose,65-99 mg/dL;Fasting Serum Glucose,65-99 mg/dL;Total Protein, 6.0-8.5 g/dL;Albumin,3.5-5.5 g/dL;Urine Protein,>=4;Urine Glucose,>=4;Urine Blood,>=4;Urine Red Blood Cells>=4;Urine White Blood Cells,>=4.
Time Frame: Period C (Day 282 to end of study)
Population: All treated participants in Period C evaluated for a specific analyte.
Measure: Number; unit: participants
Arm/Group | Abatacept (All Participants in Period C)
Number analyzed (Participants) | 153
participants
  Hemoglobin (Low) n=153 | 12
  Hematocrit (Low) n=153 | 8
  Erythrocytes (Low) n=153 | 4
  Platelet Count (Low) n=153 | 4
  Platelet Count (High) n=153 | 5
  Leukocytes (Low) n=153 | 20
  Leukocytes (High) n=153 | 18
  Absolute Neutrophils + Bands (Low) | 14
  Absolute Lymphocytes (Low) n=153 | 21
  Absolute Lymphocytes (High) n=153 | 5
  Absolute Eosinophils (High) n=153 | 50
  Alkaline Phosphatase (ALP, High) n=153 | 2
  Aspartate Aminotransferase (AST, High) | 5
  Alanine Aminotransferase (ALT, High) n=153 | 11
  G-Glutamyl Transferase (GGT, High) n=153 | 6
  Bilirubin (Total, High) n=153 | 3
  Blood Urea Nitrogen (High) n=153 | 15
  Creatinine (High) n=153 | 36
  Potassium (High) n=153 | 10
  Inorganic Phosphorus (High) n=153 | 4
  Serum Glucose (Low) n=153 | 54
  Serum Glucose (High) n=153 | 1
  Fasting Serum Glucose (Low) n=100 | 11
  Fasting Serum Glucose (High) n=100 | 7
  Total Protein (Low) n=153 | 1
  Total Protein (High) n=153 | 1
  Albumin (Low) n=153 | 9
  Urine Protein (High) n=153 | 35
  Urine Glucose (High) n=153 | 1
  Urine Blood (High) n=153 | 73
  Urine White Blood Cells (High) n=117 | 49
  Urine Red Blood Cells (High) n=117 | 86

15. Secondary Outcome: Number of Participants With Anti-Abatacept or Anti-CTLA4 Positive Responses Over Time During Open-Label Phase (Period C)
Description: During Period C, blood samples for immunogenicity assessments were obtained just prior to the start of the IV infusion of abatacept at 3-month intervals during the first 2 years of Period C, at 6-month intervals thereafter, and again 28, 56, and 85 days after the last infusion. Direct-format, enzyme-linked immunosorbent assays (ELISAs) were used to evaluate the cytotoxic T-lymphocyte antigen 4 (CTLA4) and the anti-CTLA4-T antibody.
Time Frame: Period C (Day 282 to 85 days after the last dose of study medication)
Population: All treated participants who were evaluated for immunogenicity during Period C
Measure: Number; unit: participants
Arm/Group | Abatacept (Period A Non-Responders in Period C) | Abatacept (Period C) | Placebo (Period B) to Abatacept (Period C)
Number analyzed (Participants) | 33 | 57 | 58
participants
  Anti-Abatacept, Overall on Treatment (n=31,54,54) | 1 | 5 | 2
  Anti-Abatacept, Post-Treatment (n=25,41,38) | 0 | 3 | 3
  Anti-CTLA4-T, Overall on Treatment (n=33,57,58) | 4 | 4 | 4
  Anti-CTLA4-T, Overall Post-Treatment (n=27,46,42) | 4 | 1 | 1

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 56 days up to end of study (November 2011)
Description: Study initiated: February 2004; Study completed: November 2011
Groups:
- Abatacept (Only Period A): Participants treated in Period A but did not in Periods B or C.
  Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every 2 weeks for 3 doses.
- Abatacept (Period A/Period C): Participants treated in Period A, not eligible to continue into Period B, but re-entered in Period C.
  Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every two weeks for three doses (Period A) and once a month for up to 5 years (Period C).
- Abatacept (Period A/Period B): All participants treated with Abatacept in Periods A and B who may or may not have entered Period C.
  Abatacept: 10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once every 2 weeks for 3 doses, then once a month for 6 months. If participants entered Period C, treatment continued once a month for up to 5 years.
- Abatacept (Period A)/Placebo (Period B): All participants treated with Abatacept in Period A, placebo in Period B, who may or may not have entered Period C.
  Placebo: Dextrose 5% in water (D5W) or normal saline (NS) IV infusion, once every 2 weeks for 3 doses, then monthly up to 6 months. Participants were seated or in supine position during infusion. If participants entered Period C, they were treated with Abatacept,10 milligram per kilogram body weight (mg/kg), limited to a maximum 1000 mg for participants weighing >100kg; solution infused intravenously (IV), over 90 minutes, once a month for up to 5 years.
Arm/Group | Abatacept (Only Period A) | Abatacept (Period A/Period C) | Abatacept (Period A/Period B) | Abatacept (Period A)/Placebo (Period B)
Serious Adverse Events (participants affected / at risk) | 4/32 | 10/36 | 9/60 | 14/62
Other Adverse Events (participants affected / at risk) | 22/32 | 32/36 | 57/60 | 54/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (Only Period A) (N=32) | Abatacept (Period A/Period C) (N=36) | Abatacept (Period A/Period B) (N=60) | Abatacept (Period A)/Placebo (Period B) (N=62)
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Condition aggravated (General disorders) | 0 | 1 | 0 | 0
Encephalitis (Nervous system disorders) | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (Only Period A) (N=32) | Abatacept (Period A/Period C) (N=36) | Abatacept (Period A/Period B) (N=60) | Abatacept (Period A)/Placebo (Period B) (N=62)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 5
Fatigue (General disorders) | 2 | 2 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 2 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 11 | 15
Haematuria (Renal and urinary disorders) | 0 | 2 | 5 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 8 | 8
Pharyngitis streptococcal (Infections and infestations) | 2 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 2 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 2
Vulvovaginitis (Infections and infestations) | 0 | 4 | 1 | 2
Cataract (Eye disorders) | 0 | 2 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 2 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 10 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 3 | 3 | 2
Impetigo (Infections and infestations) | 0 | 3 | 2 | 2
Pain (General disorders) | 1 | 2 | 0 | 2
Pneumonia primary atypical (Infections and infestations) | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 6 | 8 | 9
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 7 | 4
Dysuria (Renal and urinary disorders) | 0 | 0 | 4 | 4
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 4
Flushing (Vascular disorders) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 6 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 5
Tonsillitis (Infections and infestations) | 0 | 6 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 12 | 11 | 12
Urinary tract infection (Infections and infestations) | 0 | 2 | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 6 | 8 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5 | 10 | 10
Alanine aminotransferase increased (Investigations) | 0 | 0 | 5 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 4
Eosinophilia (Blood and lymphatic system disorders) | 0 | 4 | 5 | 6
Lice infestation (Infections and infestations) | 0 | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 3 | 10 | 13
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 6 | 6 | 5
Headache (Nervous system disorders) | 7 | 10 | 14 | 11
Leukocyturia (Renal and urinary disorders) | 0 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 11 | 20 | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2
Sinusitis (Infections and infestations) | 1 | 5 | 12 | 7
Vomiting (Gastrointestinal disorders) | 2 | 7 | 9 | 13
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 3 | 3 | 2
Conjunctivitis (Eye disorders) | 0 | 4 | 5 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4 | 3
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 5
Paronychia (Infections and infestations) | 2 | 3 | 3 | 2
Tinea versicolour (Infections and infestations) | 0 | 1 | 3 | 1
Varicella (Infections and infestations) | 0 | 1 | 3 | 3
Viral infection (Infections and infestations) | 3 | 0 | 2 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 8 | 4
Chills (General disorders) | 0 | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 5
Influenza (Infections and infestations) | 1 | 6 | 16 | 12
Influenza like illness (General disorders) | 0 | 0 | 3 | 4
Nausea (Gastrointestinal disorders) | 6 | 5 | 9 | 12
Otitis media acute (Infections and infestations) | 0 | 2 | 1 | 3
Pyrexia (General disorders) | 2 | 8 | 12 | 12
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less